CLINICAL TRIAL: NCT00284453
Title: Gene Expression in ICD Patients With Electrical Storm
Brief Title: Ventricular Tachyarrhythmia (VT) Storm, Gene Expression in Implantable Cardioverter Defibrillator (ICD) Patients With Electrical Storm
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sandeep Jain, MD, Assistant Professor, UPMC Heart and Vascular Institute, Cardiac Electrophysiology, University of Pittsburgh
Other Study IDs: 0510087
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmias
Keywords: ventricular; arrhythmias; ICD; VT storm; ICD patients with VT storm
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 6 RNA samples are obtained and kept frozen on-site to be evalauted at a later date. A portion of this DNA will be used to analyze the structure of certain genes that are known to play a role in cardiac arrhythmias. We cannot at this time know exatly what genes will be tested.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Forty(40)subjects that have received >2 appropriate ICD shock therapies
  Interventions: Procedure: Peripheral blood sampling
- 2: Twenty(20)subjects that have received 1-2(low level)appropriate ICD therapies
  Interventions: Procedure: Peripheral blood sampling
- 3: Ten(10)subjects that received inappropriate therapies from their ICD
  Interventions: Procedure: Peripheral blood sampling

INTERVENTIONS:
Procedure: Peripheral blood sampling — blood samples will be collected within 72 hours of subjects receiving >2, 1-2(low level) or inappropriate therapies, device data and repeat bloodwork in 3 months(+/- 4weeks).

SUMMARY:
The purpose of the proposed pilot study is to identify factors which are associated with periods of high ventricular arrhythmia burden. This will be performed by analysis of gene expression from peripheral blood samples.

DETAILED DESCRIPTION:
This is a study of patients with ICD implants who present with multiple(>2), low-level(1-2) or inappropriate therapies to their defibrillator. The purpose of this pilot study is to identify factors which are associated with periods of high ventricular arrhythmia burden by looking at gene expression from peripheral blood, in addition to levels of known markers of CHF, including catecholamine levels, B-type natriuretic peptide, and troponin. This study hypothesizes that extrinsic or systemic factors play a role in triggering these events, and if true should yield candidate proteins which would spawn functional studies to prove a role in causation. Additionally, identification of a marker of increased recurrence of events may aid in guiding therapy (starting an anti-arrhythmic versus awaiting the next event).

ELIGIBILITY:
Inclusion Criteria:

* ICD patients at least 18 years of age that present within a 72 hour period: 1) > 2 therapies for ventricular arrhythmias; 2) 1-2 therapies for ventricular arrhythmias; 3) inappropriate therapies for ventricular arrhythmias
* Able to give informed consent

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty men and women over age 18 with electrical strom that we hope will volunteer to participate in this genetic research study
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-08-26 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Genetic Testing | Day 1 Enrollment
  Identification of factors which are associated with periods of high ventricular arrhythmia burden (Day 1) by looking at gene expression from peripheral blood, in addition to levels of known markers of congestive heart failure (catecholamine levels, B-type natriuretic peptide, and troponin)in comparison to subject's return to own normal state (3 month +/- 30 days)
Genetic Testing | Day 90 +/- 30 days
  Identification of factors which are associated with periods of high ventricular arrhythmia burden (Day 1) by looking at gene expression from peripheral blood, in addition to levels of known markers of congestive heart failure (catecholamine levels, B-type natriuretic peptide, and troponin)in comparison to subject's return to own normal state (3 month +/- 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep K. Jain, M.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania